CLINICAL TRIAL: NCT04821518
Title: The Use of Samsung Health and ECG M-Trace Base II Applications for the Assessment of Exercise Tolerance as the Secondary Prevention in Patients After Brain Stroke
Brief Title: The Use of Samsung Health and ECG M-Trace Base II Applications in the Secondary Prevention After Stroke
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 1/2021
Record Dates: First submitted 2021-03-08; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Mobile Applications; Secondary Prevention; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The study group (post-stroke): The study group consisted of 26 patients in whom ischaemic brain stroke occurred within 14 days before the admission to the Clinical Department, and were hospitalised at the Department of Neurological Rehabilitation of the Clinical Department of Rehabilitation in the Wiktor Dega Orthopaedic and Rehabilitation Clinical Hospital in Poznań
- The control group: The control group was composed of 26 healthy individuals recruited from the hospital staff who did not experience stroke.

SUMMARY:
The aim of the present study was to quantitatively assess the risk factors that may affect the re-occurrence of a CVD event and the use of a commercially available mobile application Samsung Health for the assessment of parameters of exercise tolerance and the ECG M-Trace Base II application for the assessment of cardiological parameters.

DETAILED DESCRIPTION:
In the post-stroke group and in the control group, SMWT (Six Minute Walk Test) and SCT( Stair Climb Test) were preceded by a 10-minute rest in sitting position. The time of test performance, the walked distance and steps made as well as the mean and maximum gait velocity and the calories burned were assessed using the above-mentioned Samsung Health application . ECG results were assessed with the use of ECG M-Trace Base II application described above. In addition, cardiological parameters such as: systolic blood pressure (SBP) and diastolic blood pressure (DBP), heart rate (HR) and arterial blood saturation were assessed. The measurements were performed at rest and directly after SCMT and SCT. Additionally, after the tests, the level of dyspnoea and fatigue was assessed according to the modified Borg scale (score 0-10).

ELIGIBILITY:
Inclusion criteria to the post-stroke group were as follows :

1. occurrence of hemiparesis after the first episode of ischaemic stroke
2. stroke confirmed in the diagnostic imaging records
3. score >3 on Lovett's scale of muscle strength in the paretic limbs
4. score above 15 in Barthel's scale of performance in activities of daily living
5. score below 12 in the National Institutes of Health Stroke Scale (NIHSS)
6. available complete medical records concerning the assessed risk factors of recurrent CVD event
7. lack of concomitant pulmonary diseases including chronic obstructive pulmonary disease and bronchial asthma

Exclusion criteria from the post-stroke group were as follows:

1. hemiparesis or tetraparesis following many episodes of stroke,
2. lack of diagnostic imaging scans confirming the occurrence of stroke
3. hospital stay at the Department of Neurological Rehabilitation for more than 14 days from the occurrence of stroke
4. incomplete medical records concerning the assessed risk factors of recurrent CVD event
5. score >3 on Lovett's scale of muscle strength in the paretic limbs
6. score below 14 in Barthel's scale of performance in activities of daily living
7. score above 13 in the NIHSS scale
8. occurrence of factors limiting walking ability, such as diagnosed pulmonary diseases, unstable angina, severe valvular heart diseases, cardiomyopathy, musculoskeletal or autoimmune diseases.

Ages: 42 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group (post-stroke) consisted of 26 patients (mean age 54.9±7.1) in whom ischaemic stroke occurred within 14 days before the admission to the Clinical Department.
  The control group was composed of 26 healthy (mean age 55.6±6.1) individuals recruited from the hospital staff who did not experience stroke.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
heart rate at rest | baseline
  heart rate per minute
heart rate at rest | 3 weeks
  heart rate per minute
heart rate after SMWT | baseline
  heart rate per minute
heart rate after SMWT | 3 weeks
  heart rate per minute
heart rate after SCT | baseline
  heart rate per minute
heart rate after SCT | 3 weeks
  heart rate per minute
heart rhythm at rest | baseline
  heart rhythm interpreting ECG (regular or irregular)
heart rhythm at rest | 3 weeks
  heart rhythm interpreting ECG (regular or irregular)
heart rhythm after SMWT | baseline
  heart rhythm interpreting ECG (regular or irregular)
heart rhythm after SMWT | 3 weeks
  heart rhythm interpreting ECG (regular or irregular)
heart rhythm after SCT | baseline
  heart rhythm interpreting ECG (regular or irregular)
heart rhythm after SCT | 3 weeks
  heart rhythm interpreting ECG (regular or irregular)
increased blood pressure at rest | baseline
  blood pressure value [mm/Hg]
increased blood pressure at rest | 3 weeks
  blood pressure value [mm/Hg]
increased blood pressure after SMWT | baseline
  blood pressure value [mm/Hg]
increased blood pressure after SMWT | 3 weeks
  blood pressure value [mm/Hg]
increased blood pressure after SCT | baseline
  blood pressure value [mm/Hg]
increased blood pressure after SCT | 3 weeks
  blood pressure value [mm/Hg]
Distance of walk after SMWT | baseline
  Distance (metres)
Distance of walk after SMWT | 3 weeks
  Distance (metres)
Distance of walk after SCT | baseline
  Distance (metres)
Distance of walk after SCT | 3 weeks
  Distance (metres)
Steps after SMWT | baseline
  Number of steps (number)
Steps after SMWT | 3 weeks
  Number of steps (number)
Steps after SCT | baseline
  Number of steps (number)
Steps after SCT | 3 weeks
  Number of steps (number)
Velocity of walk after SMWT | baseline
  Mean velocity (km/h)
Velocity of walk after SMWT | 3 weeks
  Mean velocity (km/h)
Velocity of walk after SCT | baseline
  Mean velocity (km/h)
Velocity of walk after SCT | 3 weeks
  Mean velocity (km/h)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Chlebuś, Principal Investigator — Clinic Rehabilitation, University of Medical Sciences in Poznań
Locations (1):
- Department of Rehabilitation and Physiotherapy Rehabilitation,, Poznan, Poland

REFERENCES:
- [Derived] Lucki M, Chlebus E, Warenczak A, Lisinski P. The Use of Samsung Health and ECG M-Trace Base II Applications for the Assessment of Exercise Tolerance in the Secondary Prevention in Patients after Ischemic Stroke. Int J Environ Res Public Health. 2021 May 27;18(11):5753. doi: 10.3390/ijerph18115753. PMID 34071967